CLINICAL TRIAL: NCT07193056
Title: Chronic Kidney Disease -Mineral and Bone Disorder, The CPH-MBD Cohort
Brief Title: The CPH-MBD Cohort
Status: Not yet recruiting | Type: Observational
Sponsor: Herlev Hospital (Other)
Responsible Party: Principal Investigator, Freja Stæhr Hassager, Medical doctor, Herlev and Gentofte Hospital
Other Study IDs: H-25039131
Record Dates: First submitted 2025-09-17; First posted 2025-09-25 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Chronic Kidney Disease Mineral and Bone Disorder; Chronic Kidney Disease (CKD); Bone Markers
Keywords: bone markers; parathyroid hormone; fracture risk; bone turnover; dietary assessment
MeSH Terms: conditions — Chronic Kidney Disease-Mineral and Bone Disorder; Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 25 Years
Biospecimen Retention: Samples Without DNA — Urine, plasma and serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CPH-MBD cohort: Participants will be followed-up for 25 years after inclusion. Bone fractures, cardiovascular events, progression of kidney disease, end-stage kidney disease and death will be collected through linkage with registries during follow-up.
  There is no intervention in this study.
- Detailed dietary assessment: From the CPH-MBD cohort we invite 50 participants to complete a dietary assessment to obtain more accurate information about their calcium and phosphate intake.

SUMMARY:
Persons with chronic kidney disease (CKD) have a 3-fold increased risk of bone fracture and a 10-fold increased risk of cardiovascular disease than the general population. These increased risks are related to the disturbances in the mineral metabolism, and this clinical entity is termed Chronic Kidney Disease - Mineral and Bone Disorder (CKD-MBD).

The overall aim of the present project is to explore factors that may predict or associate with the development of bone and cardiovascular disease in patients with CKD and hopefully provide insight into underlying mechanisms and pathophysiological pathways for future treatment and prevention.

In a sub study investigators aim to explore the calcium and phosphate balance in patients with CKD and describe how these associate with each other as well as with kidney function (eGFR).

DETAILED DESCRIPTION:
Chronic kidney disease (CKD) is a chronic condition where the excretory kidney function (estimated glomerular filtration rate (eGFR)) is reduced and/or markers of kidney damage is present (often presented as albuminuria). CKD is classified into stages CKD G1-5 according the severity of the reduction in eGFR.

The prevalence of CKD is increasing world-wide, partly explained by the increase in the ageing population and prevalence of diabetes3. In Denmark, the prevalence of CKD in the population is 4-8% depending on the applied algorithm. CKD is a devastating disease both due to the risk of kidney failure and thereby the need for dialysis or transplantation, but also because the presence of CKD increases the risk of bone fracture, cardiovascular disease and mortality.

Disturbances in the mineral metabolism, including hyperphosphatemia and hyperparathyroidism develops as kidney function declines. These disturbances are closely related to the increased risk of bone and cardiovascular disease, and this relation has been gathered since 2009 in the clinical entity named Chronic Kidney Disease-Mineral and Bone Disorder (CKD-MBD).

The bone pathology in patients with CKD, named renal osteodystrophy, can be classified by the TMV classification. The TMV classification describes the bone Turnover, the bone Mineralization and the bone Volume, which may all be disturbed in renal osteodystrophy.

Per see, disturbances in the bone pathology, especially in the bone turnover is considered harmful to the bone strength. However, no studies have addressed if disturbances in the bone turnover increases the risk of bone fracture. This is the primary aim of the present study.

The golden standard for description of bone turnover is a bone biopsy. However, bone turnover markers may describe the bone turnover with a reasonable validity, and will be used in the present study to describe the turnover, as bone biopsy is not considered feasible in 1000 patients.

Especially, the low bone turnover has been a frightened condition as former studies have found an association between low bone turnover and progression of vascular calcification. However, these were executed when treatment with active vitamin D and calcium were more aggressive than today. Treatments that may also affect the vascular calcification. Therefore, it is uncertain if low bone turnover predicts cardiovascular disease. This will also be explored in the present study.

Bone and cardiovascular disease often co-occur in patients with CKD. Preclinical and clinical studies has suggested a bone vascular tissue crosstalk in CKD that may be a mediator of the high risk of fracture and cardiovascular events in patients with CKD. In the present study, it will be possible to explore how these factors, including sclerostin, Dkk-1, and Activin A, associate with changes in bone mineral density (BMD) and future fracture and cardiovascular disease.

Sarcopenia is an age-related disease characterized by a progressive decline in muscle function and mass. Sarcopenia is associated with numerous adverse health outcomes in the general population, including increased risk of falls, fractures, and mortality. Low BMD predicts an increased risk of fracture in the general population as well as in patients with CKD. A few studies have found an association between osteoporosis and sarcopenia in patients with CKD. This association between bone fragility and sarcopenia may be due to common risk factors such as age, sex, and malnutrition, but increasing evidence points towards an interaction between muscles and bone, giving rise to the uniting term osteosarcopenia. The present study will explore if sarcopenia predicts decline in BMD and future fracture.

Patients with CKD are often put on a strict diet to reduce their intake of phosphorous, potassium, sodium and protein. In theory, these dietary restrictions may in turn cause malnutrition, sarcopenia and increased risk of fall and fracture. Especially, the reduced calcium intake due to phosphorous restriction have been speculated to impact on the bone quality. This study will determine the habitual dietary intake of phosphate and calcium in patients with CKD4-5 and explore the association with bone quantity and sarcopenia.

A novel urine acid/base-score (calculated on the basis of urine pH and urine ammonium) assesses the renal tubular capacity for acid excretion and the degree of subclinical acid retention. This disease marker has been found to be largely independent of traditional kidney disease markers and robustly associated with CKD progression and incident ESKD in CKD stage 3-4 patients. This study will determine the association between the subclinical acid retention and clinical outcomes.

The study will include 1000 patients with chronic kidney disease. The patients will be recruited from the outpatient clinic at the Department of Nephrology at Herlev Hospital. The sub study focused on calcium and phosphate balance will include 50 patients with chronic kidney disease.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* CKD stage 4-5nonD (eGFR ≤ 29 ml/min) according to KDIGO (Kidney Disease Improving Global Outcome) definition

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited from the outpatient clinic, Department of Nephrology at Herlev Hospital. The outpatient clinic has approximately 1500 patients with CKD4-5nonD.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2055-01 (Estimated); Study Completion 2055-01 (Estimated)

PRIMARY OUTCOMES:
Difference in time to first fracture between patients with normal bone turnover and low bone turnover based on bone turnover markers at baseline | 25 years

SECONDARY OUTCOMES:
Time to fracture | 25 years
  All patients will be followed-up and fractures will be registered
Time to cardiovascular event | 25 years
  All patients will be followed-up and cardiovascular events will be registered
Progression in kidney disease | 25 years
  All patients will be followed-up and kidney function will be registered
Time to end-stage kidney disease | 25 years
  All patients will be followed-up and need for dialysis/kidney transplant will be registered.
Time to death | 25 years
  All patients will be followed-up and death will be registered.
Intake of calcium | Daily (for the first three days after inclusion)
  Photos of meals and written description
Intake of phosphate | Daily (for the first three days after inclusion)
  Photos of meals and written description

CONTACTS AND LOCATIONS:
Overall Officials: Ditte Hansen, Medical doctor, professor, Study Director — Department of Nephrology, Herlev Hospital

IPD SHARING:
Plan to Share IPD: No
We do not plan to share IPD as the trial will be conducted according to local legislation (Databeskyttelsesloven, Databeskyttelsesforordningen and Sundhedsloven), which does not allow sharing data.

REFERENCES:
- [Background] Naylor KL, McArthur E, Leslie WD, Fraser LA, Jamal SA, Cadarette SM, Pouget JG, Lok CE, Hodsman AB, Adachi JD, Garg AX. The three-year incidence of fracture in chronic kidney disease. Kidney Int. 2014 Oct;86(4):810-8. doi: 10.1038/ki.2013.547. Epub 2014 Jan 15. PMID 24429401
- [Background] Stevens PE, Levin A; Kidney Disease: Improving Global Outcomes Chronic Kidney Disease Guideline Development Work Group Members. Evaluation and management of chronic kidney disease: synopsis of the kidney disease: improving global outcomes 2012 clinical practice guideline. Ann Intern Med. 2013 Jun 4;158(11):825-30. doi: 10.7326/0003-4819-158-11-201306040-00007. PMID 23732715
- [Background] Svendsen SL, Rousing AQ, Carlsen RK, Khatir D, Jensen D, Hansen NM, Salomo L, Birn H, Buus NH, Leipziger J, Sorensen MV, Berg P. A Urine pH-Ammonium Acid/Base Score and CKD Progression. J Am Soc Nephrol. 2024 Nov 1;35(11):1533-1545. doi: 10.1681/ASN.0000000000000447. Epub 2024 Jul 17. PMID 39485702
- [Background] Evenepoel P, Jorgensen HS, Bover J, Davenport A, Bacchetta J, Haarhaus M, Hansen D, Gracia-Iguacel C, Ketteler M, McAlister L, White E, Mazzaferro S, Vervloet M, Shroff R. Recommended calcium intake in adults and children with chronic kidney disease-a European consensus statement. Nephrol Dial Transplant. 2024 Jan 31;39(2):341-366. doi: 10.1093/ndt/gfad185. PMID 37697718
- [Background] Moretti A, Iolascon G. Sclerostin: clinical insights in muscle-bone crosstalk. J Int Med Res. 2023 Aug;51(8):3000605231193293. doi: 10.1177/03000605231193293. PMID 37632438
- [Background] Li G, Zhang L, Wang D, AIQudsy L, Jiang JX, Xu H, Shang P. Muscle-bone crosstalk and potential therapies for sarco-osteoporosis. J Cell Biochem. 2019 Sep;120(9):14262-14273. doi: 10.1002/jcb.28946. Epub 2019 May 20. PMID 31106446
- [Background] Iwasaki Y, Kazama JJ, Fukagawa M. Molecular Abnormalities Underlying Bone Fragility in Chronic Kidney Disease. Biomed Res Int. 2017;2017:3485785. doi: 10.1155/2017/3485785. Epub 2017 Mar 22. PMID 28421193
- [Background] Rashid A, Chaudhary Hauge S, Suetta C, Hansen D. "Sarcopenia and risk of osteoporosis, falls and bone fractures in patients with chronic kidney disease: A systematic review". PLoS One. 2022 Jan 21;17(1):e0262572. doi: 10.1371/journal.pone.0262572. eCollection 2022. PMID 35061818
- [Background] Lai S, Muscaritoli M, Andreozzi P, Sgreccia A, De Leo S, Mazzaferro S, Mitterhofer AP, Pasquali M, Protopapa P, Spagnoli A, Amabile MI, Molfino A. Sarcopenia and cardiovascular risk indices in patients with chronic kidney disease on conservative and replacement therapy. Nutrition. 2019 Jun;62:108-114. doi: 10.1016/j.nut.2018.12.005. Epub 2018 Dec 11. PMID 30875540
- [Background] Cruz-Jentoft AJ, Bahat G, Bauer J, Boirie Y, Bruyere O, Cederholm T, Cooper C, Landi F, Rolland Y, Sayer AA, Schneider SM, Sieber CC, Topinkova E, Vandewoude M, Visser M, Zamboni M; Writing Group for the European Working Group on Sarcopenia in Older People 2 (EWGSOP2), and the Extended Group for EWGSOP2. Sarcopenia: revised European consensus on definition and diagnosis. Age Ageing. 2019 Jul 1;48(4):601. doi: 10.1093/ageing/afz046. No abstract available. PMID 31081853
- [Background] Mace ML, Egstrand S, Morevati M, Olgaard K, Lewin E. New Insights to the Crosstalk between Vascular and Bone Tissue in Chronic Kidney Disease-Mineral and Bone Disorder. Metabolites. 2021 Dec 7;11(12):849. doi: 10.3390/metabo11120849. PMID 34940607
- [Background] Mace ML, Gravesen E, Nordholm A, Egstrand S, Morevati M, Olgaard K, Lewin E. The Calcified Vasculature in Chronic Kidney Disease Secretes Factors that Inhibit Bone Mineralization. JBMR Plus. 2022 Mar 1;6(4):e10610. doi: 10.1002/jbm4.10610. eCollection 2022 Apr. PMID 35434452
- [Background] Barreto DV, Barreto Fde C, Carvalho AB, Cuppari L, Draibe SA, Dalboni MA, Moyses RM, Neves KR, Jorgetti V, Miname M, Santos RD, Canziani ME. Association of changes in bone remodeling and coronary calcification in hemodialysis patients: a prospective study. Am J Kidney Dis. 2008 Dec;52(6):1139-50. doi: 10.1053/j.ajkd.2008.06.024. Epub 2008 Sep 27. PMID 18824289
- [Background] Jorgensen HS, Behets G, Viaene L, Bammens B, Claes K, Meijers B, Naesens M, Sprangers B, Kuypers D, Cavalier E, D'Haese P, Evenepoel P. Diagnostic Accuracy of Noninvasive Bone Turnover Markers in Renal Osteodystrophy. Am J Kidney Dis. 2022 May;79(5):667-676.e1. doi: 10.1053/j.ajkd.2021.07.027. Epub 2021 Oct 26. PMID 34710517
- [Background] Salam S, Gallagher O, Gossiel F, Paggiosi M, Khwaja A, Eastell R. Diagnostic Accuracy of Biomarkers and Imaging for Bone Turnover in Renal Osteodystrophy. J Am Soc Nephrol. 2018 May;29(5):1557-1565. doi: 10.1681/ASN.2017050584. Epub 2018 Mar 19. PMID 29555831
- [Background] Haarhaus M, Evenepoel P; European Renal Osteodystrophy (EUROD) workgroup; Chronic Kidney Disease Mineral and Bone Disorder (CKD-MBD) working group of the European Renal Association-European Dialysis and Transplant Association (ERA-EDTA). Differentiating the causes of adynamic bone in advanced chronic kidney disease informs osteoporosis treatment. Kidney Int. 2021 Sep;100(3):546-558. doi: 10.1016/j.kint.2021.04.043. Epub 2021 Jun 5. PMID 34102219
- [Background] Moe S, Drueke T, Cunningham J, Goodman W, Martin K, Olgaard K, Ott S, Sprague S, Lameire N, Eknoyan G; Kidney Disease: Improving Global Outcomes (KDIGO). Definition, evaluation, and classification of renal osteodystrophy: a position statement from Kidney Disease: Improving Global Outcomes (KDIGO). Kidney Int. 2006 Jun;69(11):1945-53. doi: 10.1038/sj.ki.5000414. PMID 16641930
- [Background] Kidney Disease: Improving Global Outcomes (KDIGO) CKD-MBD Update Work Group. KDIGO 2017 Clinical Practice Guideline Update for the Diagnosis, Evaluation, Prevention, and Treatment of Chronic Kidney Disease-Mineral and Bone Disorder (CKD-MBD). Kidney Int Suppl (2011). 2017 Jul;7(1):1-59. doi: 10.1016/j.kisu.2017.04.001. Epub 2017 Jun 21. No abstract available. PMID 30675420
- [Background] Vestergaard SV, Christiansen CF, Thomsen RW, Birn H, Heide-Jorgensen U. Identification of Patients with CKD in Medical Databases: A Comparison of Different Algorithms. Clin J Am Soc Nephrol. 2021 Apr 7;16(4):543-551. doi: 10.2215/CJN.15691020. Epub 2021 Mar 11. PMID 33707181
- [Background] Xie Y, Bowe B, Mokdad AH, Xian H, Yan Y, Li T, Maddukuri G, Tsai CY, Floyd T, Al-Aly Z. Analysis of the Global Burden of Disease study highlights the global, regional, and national trends of chronic kidney disease epidemiology from 1990 to 2016. Kidney Int. 2018 Sep;94(3):567-581. doi: 10.1016/j.kint.2018.04.011. Epub 2018 Aug 3. PMID 30078514
- [Background] Kidney Disease: Improving Global Outcomes (KDIGO) CKD-MBD Work Group. KDIGO clinical practice guideline for the diagnosis, evaluation, prevention, and treatment of Chronic Kidney Disease-Mineral and Bone Disorder (CKD-MBD). Kidney Int Suppl. 2009 Aug;(113):S1-130. doi: 10.1038/ki.2009.188. PMID 19644521

DOCUMENTS (1):
  • Study Protocol (2025-09-26): https://cdn.clinicaltrials.gov/large-docs/56/NCT07193056/Prot_001.pdf